CLINICAL TRIAL: NCT04895332
Title: BPOI (Berlin Pediatric Oxygenation Index) - A New Predictor for Imminent Failure of HFNC in Children Avoiding Delayed NIV or Intubation
Status: Withdrawn | Type: Observational
Why Stopped: Due to pandemia
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Department of Anesthesiology and Operative Intensive Care Medicine (CCM/CVK), Charite University, Berlin, Germany
Other Study IDs: BPOI
Record Dates: First submitted 2021-05-17; First posted 2021-05-20 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Respiratory Failure (Pediatric Patients)
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators developed an index that integrates different flow-settings in High-flow nasal cannula (HFNC) therapy with non-invasively measured clinical parameters of oxygenation in pediatric patients. This observational study is designed to evaluate this index and to determine a cut-off value for imminent HFNC failure.

DETAILED DESCRIPTION:
High-flow nasal cannula therapy is a broadly used instrument of respiratory support in pediatric and adult patients with respiratory failure.

For adult patients with pneumonia and respiratory failure, there is a validated index (ROX; ratio SpO2/FiO2) which helps to identify those at risks for the need of intubation.

This index however is not applicable in the pediatric population because the physiological values of respiratory rate vary greatly across different ages.

Thus, based on the particularities of pediatric patients the investigators developed an index that integrates different flow-settings in HFNC therapy with non-invasively measured clinical parameters of oxygenation. The BPOI is defined as the ratio of the product of the peripherally measured oxygen saturation and the patient's body weight divided by the product of HFNC flow and the fraction of inspired oxygen:

BPOI = (SpO2 * kg) / (Flow * FiO2)

ELIGIBILITY:
Inclusion Criteria:

* Patients with respiratory failure and indication für High-flow nasal cannula therapy
* Patients aged between 4 1/7 weeks and 18 years
* Patients who were treated between 01/01/2017 and 28/02/2021 in the Department of Pediatric Pulmonology, Immunology and Intensive Care Medicine at Campus Virchow- Klinikum, Charité - Universitätsmedizin Berlin

Exclusion Criteria:

* Patients aged between 1 and 27 days (neonatal period)
* Patients with congenital cyanotic heart defects
* Patients after or in the course of haematopoetic stem cell transplantation
* Patients with ambulatory respiratory support

Ages: 28 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric Patients with respiratory failure and High-flow nasal cannula therapy (HFNC).
  Approximately 220 patients will be enrolled in the observational study. Their data collected during their entire hospital stay which is saved on the clinical data processing system will be evaluated to reproduce the BPOI (BPOI = (SpO2 * kg) / (Flow * FiO2) ) We will compare the indices of patients who failed and those who were successfully treated with HFNC therapy. Failure is defined by the need for non-invasive or invasive mechanical ventilation.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
BPOI (Berlin Pediatric Oxygenation Index) | 01.01.2017-28.02.2021
  Evaluation of a certain cut-off value for the BPOI (Berlin Pediatric Oxygenation Index) that predicts imminent failure of high-flow nasal cannula (HFNC) therapy in paediatric patients.

SECONDARY OUTCOMES:
Heart rate | 01.01.2017-28.02.2021
  Measurement of heart rate at given time points
Respiratory rate | 01.01.2017-28.02.2021
  Measurement of respiratory rate at given time points
Blood pressure (mean arterial pressure, MAP) | 01.01.2017-28.02.2021
  Measurement of blood pressure at given time points
Intensive care unit length of stay | 01.01.2017-28.02.2021
  Time period until the patient is either deferred to another non-ICU or until end of treatment period/death
High-flow nasal cannula therapy failure | 01.01.2017-28.02.2021
  Count of days until the respiratory therapy is escalated to non-invasive ventilation after the cut-off value for the BPOI has been reached.
Need for intubation | 01.01.2017-28.02.2021
  High-flow nasal cannula (HFNC) or non-invasively ventilation (NIV failure)
Need for mechanical ventilation | 01.01.2017-28.02.2021
  Need for assisted or controlled ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Charite University, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No